CLINICAL TRIAL: NCT00002860
Title: A Phase II Trial of Complete Surgical Resection For Stage IV Melanoma -- Surgical Resection With Biological Evaluation and Clinical Follow-Up
Brief Title: SWOG-9430: Surgery in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065130; U10CA032102 (NIH); SWOG-9430; ECOG-S9430
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery (Other)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Complete surgical resection of metastatic melanoma

SUMMARY:
RATIONALE: Surgery may be effective therapy in treating patients with metastatic melanoma.

PURPOSE: This phase II trial is studying how well surgery works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess overall and progression-free survival in patients with metastatic melanoma (beyond the draining lymph nodes) after complete surgical resection of all known disease.
* Determine the ability of the Southwest Oncology Group Melanoma Committee to enroll patients with metastatic melanoma who can be resected to a disease-free state.

OUTLINE: This is a multicenter study.

All patients undergo gross total resection of all known disease. Patients whose disease cannot be completely resected or who have disease recurrence after surgery are removed from study. Patients found to have microscopic residual disease after surgery are considered completely resected. Resected tissue is submitted for analysis on protocol SWOG-9431.

Patients may receive any adjuvant therapy (e.g., radiotherapy, interferon, and/or vaccines) deemed clinically appropriate by the treating physician.

Patients are followed periodically for 5 years after study entry.

PROJECTED ACCRUAL: A total of 100 eligible patients with completely surgically resected disease will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma that is deemed grossly surgically resectable

  * Multiple resected sites or metastatic melanoma of unknown primary allowed provided all known disease can be grossly resected
  * Recurrence in iliac lymph nodes after inguinal lymph dissection allowed
* No metastatic disease beyond the lesions planned for resection

  * Confirmed by CT scan of chest, abdomen, pelvis, and CT or MRI of brain within 42 days of study
* Concurrent registration on protocol SWOG-9431 required

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer from which patient is currently disease free
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior immunotherapy in the adjuvant or metastatic setting allowed

Chemotherapy:

* Prior chemotherapy in the adjuvant or metastatic setting allowed

Endocrine therapy:

* Prior hormonal therapy in the adjuvant or metastatic setting allowed

Radiotherapy:

* Prior radiotherapy in the adjuvant or metastatic setting allowed

Surgery:

* See Disease Characteristics
* At least 14 days since prior surgery in the adjuvant or metastatic setting

Other:

* Recovered from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 1996-11; Primary Completion 2006-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Sosman, MD, Study Chair — Vanderbilt-Ingram Cancer Center; John M. Kirkwood, MD, Study Chair — University of Pittsburgh
Locations (124):
- United States (124):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Banner Thunderbird Medical Center, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Harrington Cancer Center, Amarillo, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Sondak VK, Liu PY, Warneke J, et al.: Surgical resection for stage IV melanoma: a Southwest Oncology Group trial (S9430). [Abstract] J Clin Oncol 24 (Suppl 18): A-8019, 457s, 2006.